CLINICAL TRIAL: NCT02661646
Title: Assessment of Quality of Life Changes on Lower Extremity Lymphedema Patients Using an Advanced Pneumatic Compression Device at Home
Brief Title: Quality of Life Changes on Lower Extremity Lymphedema Patients Using an Advanced Pneumatic Compression Device (PCD)
Status: Terminated | Type: Observational
Why Stopped: Due to slow enrollment during COVID
Sponsor: Tactile Medical (Industry)
Responsible Party: Sponsor
Other Study IDs: 5010
Record Dates: First submitted 2016-01-18; First posted 2016-01-22 (Estimated); Last update posted 2023-04-03 (Actual); Status verified 2023-03

CONDITIONS: Lymphedema
Keywords: Chronic Swelling; Leg Lymphedema; Primary Lymphedema; Secondary Lymphedema
MeSH Terms: conditions — Lymphedema

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Advanced Pneumatic Compression Group: All study participants will receive treatment using an advanced pneumatic compression device.
  Interventions: Device: Advanced Pneumatic Compression Device

INTERVENTIONS:
Device: Advanced Pneumatic Compression Device — Advanced Pneumatic Compression Device
  Other Names: Flexitouch system; Flexitouch Plus

SUMMARY:
Assessment of quality of life and symptoms changes in primary or secondary, unilateral or bilateral lower extremity lymphedema patients using an advanced pneumatic compression system.

DETAILED DESCRIPTION:
Post-market, on label, multi-center, single arm, observational clinical trial of a prospective cohort of 300 subjects with primary or secondary, unilateral or bilateral, lower extremity lymphedema in the United States. All subjects will receive pneumatic compression treatment for 52 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Diagnosis of primary or secondary, unilateral or bilateral, lower extremity lymphedema
* Ability and willingness to participate in all aspects of the study including following prescribed care
* Ability to provide informed consent
* Must have a prescription for the Flexitouch (Flexitouch system or Flexitouch Plus)

Exclusion Criteria:

* Diagnosis of active or recurrent cancer, or less than 3 months at the time of initial evaluation from the completion of chemotherapy, radiation therapy or primary surgery for the treatment of cancer.
* Active skin or limb infection/inflammatory disease (acute cellulitis, or other uncontrolled skin or untreated inflammatory skin disease)
* Acute thrombophlebitis (in last 2 months)
* Pulmonary embolism within the previous 6 months
* Deep Vein Thrombosis (DVT) within the previous 3 months
* Severe peripheral artery disease (critical limb ischemia including ischemic rest pain, arterial wounds, or gangrene)
* Pulmonary edema
* Heart failure (acute pulmonary edema, decompensated acute heart failure)
* Patients with poorly controlled asthma
* Previous use of the study pneumatic compression device (PCD)
* Currently using multi-layer bandaging (MLB) unless bandages can be removed for limb circumference measurements
* Pregnant women or women of childbearing potential not on contraception
* Any condition where increased venous and lymphatic return is undesirable
* Currently participating in another medical device or drug clinical trial
* Signs of noncompliance at the week 4 visit including: using the device less than 3 times per week and/or not attending the scheduled visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary or secondary, unilateral or bilateral, lower extremity lymphedema patients using the Flexitouch system during a 52 week study period.
  *Note: Only Veteran's are eligible as this study is run through The Department of Veterans Affairs New York Harbor Healthcare System.
Sampling Method: Non-Probability Sample
Enrollment: 249 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
Quality of life changes: Questionnaires | 12 weeks
  Questionnaires to assess quality of life changes after 12 weeks of treatment
Lymphedema symptom changes | 12 weeks
  Questionnaires [Lymphedema Quality of Life Tool (LYMQOL)] to assess lymphedema. symptom changes after 12 weeks of treatment. LYMQOL includes sub-scores for Function (range 8-32), Appearance (range 7-28), Symptoms (range 5-20), and Mood (range 6-24) where lower scores represent a better outcome. It also includes an Overall QOL sub-score (range 0-10) where a higher score represents a better outcome.
Number of lymphedema and venous related healthcare visits | 52 weeks
  Comparison of the number of lymphedema and venous related health care visits the year preceding treatment and the during the 52 weeks while receiving treatment (or until study exit)

SECONDARY OUTCOMES:
Limb circumference changes after 12 weeks and 52 weeks of treatment | 12 weeks and 52 weeks
  Comparison of changes in limb circumference after 12 weeks and 52 weeks of treatment
Fibrosis grading changes after 12 weeks and 52 weeks of treatment | 12 weeks and 52 weeks
  Comparison of fibrosis grading (range Grade 0 to Grade 3, a lower grade represents a better outcome) after 12 weeks and 52 weeks of treatment
Assessment of skin changes after 12 weeks and 52 weeks of treatment | 12 weeks and 52 weeks
  Comparison of changes in the presence of skin conditions based on clinician observation after 12 weeks and 52 weeks of treatment
Lymphedema staging changes after 12 weeks and 52 weeks of treatment | 12 weeks and 52 weeks
  Comparison of lymphedema staging (range Grade 0 to Grade 3, a lower grade represents a better outcome) after 12 weeks and 52 weeks of treatment
Quality of life changes: Questionnaires | 24 weeks and 52 weeks
  Questionnaires to assess quality of life changes after 24 weeks of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Maldonado, MD, Principal Investigator — NYU
Locations (6):
- United States (6):
  - VA Maryland Healthcare System, Baltimore, Maryland
  - VA New Jersey Health Care System (VANJHCS), East Orange, New Jersey
  - VA NY Harbor Healthcare System - Brooklyn, Brooklyn, New York
  - VA Western New York Healthcare System, Buffalo, New York
  - VA NY Harbor Healthcare System - St. Albans, Jamaica, New York
  - VA NY Harbor Healthcare System - Manhattan, New York, New York

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-07-03): https://cdn.clinicaltrials.gov/large-docs/46/NCT02661646/Prot_SAP_000.pdf
  • Informed Consent Form (2021-05-04): https://cdn.clinicaltrials.gov/large-docs/46/NCT02661646/ICF_001.pdf